CLINICAL TRIAL: NCT03209986
Title: Randomized Control Trial of Mesenchymal Stem Cell Transplantation in Decompensated Liver Cirrhosis Resulted From Viral Hepatitis
Brief Title: Trial of Mesenchymal Stem Cell Transplantation in Decompensated Liver Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Consultant Physician, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJMSC0001
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Liver Cirrhosis
Keywords: Liver Cirrhosis; Mesenchymal Sem Cells
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blind to the randomization results of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC group (Experimental): mesenchymal stem cell transplantation via peripheral vein: 1x10E6 MSCs/kg body weight administered via peripheral vein at week 0, 4, 8.
  Interventions: Procedure: mesenchymal stem cell transplantation via peripheral vein; Other: mesenchymal stem cell
- control (No Intervention): Standard medication for viral hepatitis and cirrhosis

INTERVENTIONS:
Procedure: mesenchymal stem cell transplantation via peripheral vein — 1x10E6 MSCs/kg body weight will be administered via peripheral vein for 3 times at week 0, 4 and 8
  Arms: MSC group
Other: mesenchymal stem cell — mesenchymal stem cell infusion produced by Cell products of National Engineering Research Center(short for CPNERC), Tianjin, China
  Arms: MSC group

SUMMARY:
There has been great interest in recent years to take advantage of stem cells to treat liver cirrhosis. Mesenchymal stem cells (MSC) has been shown to be safe and effective for liver diseases in some studies. Randomization controlled studies are needed to confirm the long term effect of MSC treatment for liver cirrhosis. This study aimed to investigate the safety and efficacy of mesenchymal stem cells in hepatitis B and C related liver cirrhosis patients.

This study is an open-label multicenter randomized control study. Patients with with decompensated cirrhosis will be randomly assigned to receive MSC treatment plus standard medical care(treatment）or standard medical care (control). Three times of MSC infusion (1x10E6 cells/kg body weight) via peripheral vein will be given to the experimental group (once in 4 weeks). The primary outcome is absolute change in liver function indexes and and scores. Secondary outcomes are cirrhosis-related complications, symptoms, life quality, and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. HBV -related liver cirrhosis
3. Child-Pugh score ≥7
4. With presentations of decompensation
5. Written consent

Exclusion Criteria:

1. Hepatocellular carcinoma or other malignancies
2. Severe problems in other vital organs(e.g.the heart,renal or lungs)
3. Pregnant or lactating women
4. Severe bacteria infection
5. Anticipated with difficulty of follow-up observation
6. Coinfection with HIV or other viral hepatitis.
7. Drug abuse or alcohol abuse
8. History of severe allergy to biological products
9. Other candidates who are judged to be not applicable to this study by doctors -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Change of liver functions as assessed by MELD score | 1 year
  Change of liver functions as assessed by MELD score (MELD, Model for End-Stage Liver Disease Score: MELD = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43)
Safety: Adverse events as assessed according to CTCAE 4.03 | 1 year
  Adverse events as assessed according to CTCAE 4.03

SECONDARY OUTCOMES:
Survival Benefit: Survival Rate at different time points | 1 year, 2 year and 5 years
  survival rate at different time points
Histological change of the liver: Histological scores assessed by liver biopsy | 1 year, 2 year and 5 years
  histological scores assessed by liver biopsy at baseline and after treatment
Clinical benefit: Incidences of cirrhosis-related complications such as GI bleeding, ascites, hepatorenal syndrome, hepatoencephalopathy | 1, 2 and 5 years
  Incidences of cirrhosis-related complications such as GI bleeding, ascites, hepatorenal syndrome, hepatoencephalopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Disease, Xijing Hospital, Xi'an, Shaanxi, China